CLINICAL TRIAL: NCT05636098
Title: Repeatability and Reproducibility of Oxygen Reserve Index (ORi)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1050
Record Dates: First submitted 2022-11-23; First posted 2022-12-05 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Masimo Rainbow Sensors (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo Rainbow Sensors.
  Interventions: Device: Masimo Rainbow Sensors

INTERVENTIONS:
Device: Masimo Rainbow Sensors — Noninvasive pulse oximeter sensor

SUMMARY:
This study is designed to evaluate the repeatability and reproducibility of ORi using an investigational Masimo rainbow sensor and FDA cleared rainbow sensors connected to the Masimo Radical-7 pulse oximeter and Masimo Root monitor in healthy volunteers as the subjects undergo a controlled hyperoxygenation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 50 years of age.
* Subject weighs a minimum of 110 lbs.
* Hemoglobin value ≥ 11 g/dL.
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* Blood Pressure: Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥ 50 mmHg, and if systolic BP is lower than 100 mmHg and/or diastolic BP is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
* CO value ≤ 3.0% FCOHb.
* Subject is able to read and communicate in English and understands the study and the risks involved

Exclusion Criteria:

* Subject has a positive hCG test.
* Subject has a BMI > 35.
* Subject has a history of fainting (vasovagal syncope), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos or piercings, and/or has any visible healing wounds that a medical professional determines may place them at an increased risk for participation. *
* Subject has known drug or alcohol abuse.
* Subject uses recreational drugs. *
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
* Subject has any history of a stroke, myocardial infarction (heart attack), and/or seizures.
* Subject has any chronic bleeding disorder (e.g., hemophilia).
* Subject has taken anticoagulant medication within the past 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS)).
* Subject has donated blood within the past 4 weeks.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome.
* Subject has any cardiac dysrhythmia (e.g., atrial fibrillation) and has not received clearance from their physician to participate. *
* Subject has a known neurological and/or psychiatric disorder (e.g., schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's disease) that interferes with the subject's level of consciousness. *
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any active signs and/or symptoms of infectious disease (e.g., Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.). *
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year, including but not limited to major dental surgery, appendectomy, plastic surgery, jaw surgery, major ENT surgery, major abdominal and/or pelvic surgery, heart surgery, or thoracic surgery. *
* Subject has symptoms of congestion, head cold, or other illnesses.
* Subject has been in a severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
* Subject has any cancer or history of cancer (not including skin cancer). *
* Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
* Subject is allergic to Lidocaine, chlorhexidine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent diabetes, or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization or had a C-section within the past 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis), exercise (working out, riding a bike, riding a skateboard, etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Masimo Rainbow Sensors
Started | 53
Completed | 29
Not Completed | 24

BASELINE CHARACTERISTICS:
Arm/Group | Masimo Rainbow Sensors
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 4
  More than one race | 1
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Repeatability of Masimo Rainbow Sensors
Description: The Repeatability of ORi for Masimo Rainbow Sensors refers to the ability of a sensor to consistently produce the same readings under similar conditions (hyperoxia level).
  1. A Repeatability Error is defined as the difference between ORi measurements from one sensor at different time points under similar operating conditions.
  2. The mean of the absolute of all the repeatability errors obtained across different conditions and sensors is represented as the Repeatability of ORi.
  3. Since ORi is a unit-less parameter, the Repeatability of ORi is also unit-less. ORi values range from 0-1, with 0 indicating normoxia while 1 indicating moderate to high hyperoxia.
Time Frame: 1-1.5 hours
Population: 2 subjects not included in analysis for device setting errors.
Measure: Mean (Full Range); unit: Mean Absolute Error (Unitless)
Arm/Group | Masimo Rainbow Sensors
Number analyzed (Participants) | 27
Mean Absolute Error (Unitless) | 0.05 [0 to 1]

2. Primary Outcome: Reproducibility of Masimo Rainbow Sensors
Description: The Reproducibility of ORi for Masimo Rainbow Sensors refers to the ability of two sensors to produce similar ORi results when measurements are taken under the same conditions (hyperoxia level).
  1. A Reproducibility Error is the difference between 2 ORi measurements obtained from each of a pair of sensors at the same time and under the same operating conditions.
  2. The mean of absolute of all the reproducibility errors are represented as the Reproducibility of ORi.
  3. Since ORi is a unit-less parameter, the Reproducibility of ORi is also unit-less. ORi values ranges from 0-1, with 0 indicating normoxia while 1 indicating moderate to high hyperoxia.
Time Frame: 1-1.5 hours
Population: 5 subjects not included in analysis due to device setting errors.
Measure: Mean (Full Range); unit: Mean Absolute Error (Unitless)
Arm/Group | Masimo Rainbow Sensors
Number analyzed (Participants) | 22
Mean Absolute Error (Unitless) | 0.07 [0 to 1]

ADVERSE EVENTS:
Time Frame: 1-3 hours
Arm/Group | Masimo Rainbow Sensors
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT05636098/Prot_SAP_000.pdf